CLINICAL TRIAL: NCT07094945
Title: The Effect of Remimazolam on Postoperative Sleep Quality of Patients Undergoing Gynecological Day Surgery
Brief Title: The Effect of Remimazolam on Postoperative Sleep Quality
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025S076
Record Dates: First submitted 2025-07-29; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gynecological Day Surgery
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Grop (Experimental): Remimazolam 0.3mg/kg for induction and 0.6-1.0 mg/kg·h for maintenance of anesthesia
  Interventions: Drug: Remimazolam
- Propofol Group (Active Comparator): Propofol 2 mg/kg for induction and 4-12 mg/kg·h for maintenance of anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam 0.3 mg/kg is slowly injected intravenously until loss of consciousness. Remimazolam 0.6-1.0 mg/kg·h is used for anesthesia maintenance.
  Arms: Remimazolam Grop
Drug: Propofol — Propofol 2 mg/kg is slowly injected intravenously until loss of consciousness. Remimazolam 4-12 mg/kg·h is used for anesthesia maintenance
  Arms: Propofol Group

SUMMARY:
A large amount of clinical evidence shows that after surgery, especially major surgery, the sleep quality of patients often drops significantly immediately, with the most obvious decline on the first night after surgery, which can last for several days to several months. Remimazolam is a new type of benzodiazepine drug and a super-short-acting GABAA receptor agonist. Compared with propofol, remimazolam can largely avoid adverse reactions such as hemodynamic fluctuations, excessive sedation and injection pain caused by propofol. It has good safety and is superior to propofol. However, there are currently only a few clinical research results regarding the impact of remimazolam on the sleep quality of patients under general anesthesia or sedation. Therefore, this study intends to observe the effect of remimazolam on the sleep quality of patients in gynecological day surgery. It is expected that by optimizing the anesthesia plan, the postoperative sleep quality of patients can be improved, and ultimately the postoperative recovery of patients can be promoted.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification grades I - II.
* BMI: 18.5-24 kg/m ².
* Be able to correctly understand and complete the assessment scale independently.
* The operation time shall not exceed one hour.
* Informed consent for this research.

Exclusion Criteria:

* PSQI > 7 points (with sleep disorders requiring medical intervention within the last month).
* Suffering from central nervous system diseases or mental disorders.
* Patients with sleep apnea syndrome or other serious respiratory diseases.
* Have functional disorders of important organs.
* Alcohol abuse or a history of opioid, benzodiazepine or other known drug abuse that may affect sleep.
* Allergic to the research medication.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Richard Campbell's Sleep Scale score | The night of the first to third postoperative day
  Range: 0 points (optimal sleep) to 10 points (optimal sleep). Direction: The higher the score, the more severe the sleep problem

SECONDARY OUTCOMES:
Blood Pressure | Before anesthesia, before the insertion of the laryngeal mask, at the beginning of the operation, at the end of the operation, and when the laryngeal mask is removed
Heart rate | Before anesthesia, before the insertion of the laryngeal mask, at the beginning of the operation, at the end of the operation, and when the laryngeal mask is removed.
Postoperative adverse reactions | 24 hours after the operation
  such as postoperative pain, nausea, vomiting, and fatigue.